CLINICAL TRIAL: NCT06954194
Title: The Efficacy of Explicit vs. Implicit Intervention Procedures for Cantonese Children With Developmental Language Disorder: A Randomized Controlled Trial
Brief Title: Syntactic Intervention for Cantonese-speaking Children With DLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, ZHANG Caicai, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20220505001-02; 20211061 (Other Grant/Funding Number: Food and Health Bureau of Hong Kong SAR)
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Developmental Language Disorder
Keywords: Randomized Controlled Trial; Explicit intervention; Implicit intervention; Procedural circuit Deficit Hypothesis; Individual difference; Relative clause; Syntactic priming; Shape coding
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Explicit intervention group (Experimental): Participants in this group will receive explicit teaching of the target structure using the Shape Coding scheme adapted to be age- and language (Cantonese)-appropriate, followed by syntactic priming sessions.
  Interventions: Behavioral: Explicit intervention (Shape Coding+syntactic priming)
- Implicit intervention group (Active Comparator): Participants in this arm will receive identical syntactic priming sessions to the explicit intervention group, but without explicit teaching of the target structure using the Shape Coding scheme.
  Interventions: Behavioral: Implicit intervention (syntactic priming only)

INTERVENTIONS:
Behavioral: Explicit intervention (Shape Coding+syntactic priming) — For explicit intervention, a syntactic priming task will be preceded by explicit teaching of the target structure using the Shape Coding scheme adapted to be age- and language (Cantonese)-appropriate. A different set of 10 sentences will be used for teaching in each explicit intervention session, with five sentences used as exemplars for the experimenter to explain the target structure, and the remaining five sentences for children to practice. The syntactic priming session will be presented as a game to sustain the children's interest and to disguise the purpose of the study. Each intervention session will contain 40 pairs of prime-target pictures, 40 pairs of control-target pictures, and 20 pairs of filler pictures, randomly presented to the experimenter and child and controlled by the experimenter. In total, there are 500 doses of SRC-O sentences (50 sentences x10 sessions).
  Arms: Explicit intervention group
Behavioral: Implicit intervention (syntactic priming only) — For implicit intervention, the same 10 sessions of syntactic priming will be provided to the children without explicit instruction of the SRC-O structure using the Shape Coding System. Nonetheless, to make the exposure and dosage as comparable as possible between the two groups, children in the implicit intervention group will also receive 10 listening sessions before the syntactic priming sessions. During the listening sessions, the same sets of sentences used in the explicit instruction sessions will be presented and the children will be instructed to listen closely as the tutor reads aloud the SRC-O sentence. Each listening session will be followed by a syntactic priming session that is identical to that of the explicit intervention group. In total, there are also 500 doses of SRC-O sentences (50 sentences x10 sessions).
  Arms: Implicit intervention group

SUMMARY:
The goal of this clinical trial is to compare the efficacy of explicit vs. implicit intervention on subject relative clause production in Cantonese-speaking children with Developmental Language Disorder (DLD). It will also learn about individual difference predictors of intervention outcomes. The main questions it aims to answer are:

1. Will the explicit intervention (Shape Coding+syntactic priming) on relative clause production lead to better outcomes than implicit intervention (syntactic priming only)?
2. Can pre-intervention procedural learning, working memory (WM) capacities, and grammar impairment severity predict the intervention outcomes across children with DLD?
3. Will 10 intervention sessions (500 doses of the target structure) lead to learning progress in children with DLD, even with implicit intervention, and will the progress plateau at some point of the intervention?

Researchers will compare the explicit intervention to the implicit intervention to see if the explicit intervention leads to better interventional outcomes.

Participants will:

* Undergo diagnostic assessments of DLD to confirm their DLD status.
* Complete pre-intervention assessments to assess their procedural learning and working memory capacities.
* Undergo the intervention phase, which consists of a pretest, 10 intervention sessions, three posttests (after the 1st, 5th and 10th intervention), and a retention test (1 month after the last intervention).

DETAILED DESCRIPTION:
This project is the first to adopt a randomized controlled trial (RCT) to compare the efficacy of explicit vs. implicit intervention on relative clause production (subject relative clause in object position of the main clause or SRC-O) in Cantonese-speaking children with DLD and to use an individual difference approach to identify predictors of intervention outcomes.

The investigators aim to examine the following three specific questions:

1. Will the explicit intervention (Shape Coding+syntactic priming) on relative clause production lead to better outcomes than implicit intervention (syntactic priming only)? Based on the Procedural circuit Deficit Hypothesis (PDH), the investigators hypothesize that explicit intervention would switch the reliance of learning to the relatively intact declarative learning circuitry and lead to better outcomes than implicit intervention.
2. Can pre-intervention procedural learning, working memory (WM) capacities, and grammar impairment severity predict the intervention outcomes across children with DLD? Based on the PDH, the investigators hypothesize that children with lower procedural learning abilities will demonstrate worse outcomes in the implicit intervention group, but better outcomes in the explicit intervention group. As for WM and grammar impairment, the investigators hypothesize that children with better WM or grammatical abilities will demonstrate better outcomes in both groups.
3. Will 10 intervention sessions (500 doses of the target structure) lead to learning progress in children with DLD, even with implicit intervention, and will the progress plateau at some point of the intervention? As informed by previous studies, the investigators hypothesize that more exposure to the target structure, especially with high variability in the input, will lead to improvement, even for the implicit intervention group. The investigators will explore whether the progress will plateau over the course of interventions and compare the learning trajectory between explicit and implicit interventions.

A total of 32 Cantonese-speaking school-age children with DLD (5-8 years old) will be recruited (N=16/group). The children will be pre-screened with an online questionnaire on language background and case history, and then assessed on the Raven's Standard Progressive Matrices (~25 min), hearing screening (~5 min) and Hong Kong Cantonese Oral Language Assessment Scale (HKCOLAS) (~90 min) to confirm DLD. Eligible children will be assigned to one of the two intervention groups following a random allocation sequence of letters "A" and "B" (e.g., ABBBA…), where A and B refer to the explicit and implicit intervention respectively, on a 1:1 allocation ratio.

The study consists of pre-intervention assessments and an intervention phase. For pre-intervention assessments, children's procedural learning, declarative learning, and working memory capacities will be assessed using the serial reaction time (SRT) task, old/new picture recognition task, and forward and backward digit span test, respectively. The purpose is to examine the predictive power of these capacities in the individual children's intervention outcomes.

The intervention phase includes a pretest, 10 intervention sessions, three posttests (after the 1st, 5th and 10th intervention), and a retention test (1 month after the last intervention). The pretest serves as a baseline; the three posttests are to assess maintenance of the target structure (SRC-O) after priming has ceased and the improvement over the course of interventions; the retention test is for assessing longer-term retention of the intervention outcomes.

The procedure of the pretest, three posttests and retention (~10 min/test) is identical, during which the children will be asked to describe 10 pictures without priming or feedback from the experimenter. Ten online intervention sessions (~45 min/session) will be administered to the children via zoom over four weeks, with 2-3 sessions per week.

For explicit intervention, a syntactic priming task will be preceded by explicit teaching of the target structure using the Shape Coding scheme adapted to be age- and language (Cantonese)-appropriate. A different set of 10 sentences will be used for teaching in each explicit intervention session, with five sentences used as exemplars for the experimenter to explain the target structure, and the remaining five sentences for children to practice. During the practice, the children will be asked to drag words into their corresponding shapes (e.g., oval for noun/noun phrase, rhombus for verb/verb phrase, and square for particle). All sentences will be constructed using the P1 Chinese character database to ensure that children can read the sentences.

The syntactic priming session will be presented as a game to sustain the children's interest and to disguise the purpose of the study. Each intervention session will contain 40 pairs of prime-target pictures, 40 pairs of control-target pictures, and 20 pairs of filler pictures, randomly presented to the experimenter and child and controlled by the experimenter. The game rule is to catch when two identical pictures are presented to the experimenter and child (i.e., fillers) by saying "Snap!". For each prime/control-target pair, the experimenter will describe a picture using the target structure - subject relative clause in object position of the main clause (SRC-O), and the child will produce a sentence based on the second picture. In total, there are 500 doses of SRC-O sentences (50 sentences x10 sessions).

For implicit intervention, the same 10 sessions of syntactic priming will be provided to the children without explicit instruction of the SRC-O structure using the Shape Coding System. Nonetheless, to make the exposure and dosage as comparable as possible between the two groups, children in the implicit intervention group will also receive 10 listening sessions before the syntactic priming sessions. During the listening sessions, the same sets of sentences used in the explicit instruction sessions will be presented and the children will be instructed to listen closely as the tutor reads aloud the SRC-O sentence. Each listening session will be followed by a syntactic priming session that is identical to that of the explicit intervention group. In total, there are also 500 doses of SRC-O sentences (50 sentences x10 sessions).

ELIGIBILITY:
Inclusion Criteria:

* being Cantonese dominant who learned Cantonese as their first language and attending Cantonese-medium primary schools.
* having normal IQ and no hearing impairment.
* scoring at least -1.25 SD below the mean in any two subtests of the Hong Kong Cantonese Oral Language Assessment Scale (a standardized language assessment tool for Hong Kong Cantonese-speaking children).

Exclusion Criteria:

* Autism Spectrum Disorder.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Production accuracy | From pretest to the retention test (1 month after all 10 intervention sessions are completed)
  Production accuracy of the target structure
Number of successful learners | From pretest to the retention test (1 month after all 10 intervention sessions are completed)
  The number of successful learners (≥80% accuracy)

CONTACTS AND LOCATIONS:
Overall Officials: Caicai Zhang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Speech and Language Sciences Laboratory (SLS Lab), Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided